CLINICAL TRIAL: NCT03973424
Title: Mobile Methods for Reducing Obesity Risk in Parents and Children: A Randomized Trial
Brief Title: Mobile Methods for Reducing Obesity Risk in Parents and Children
Acronym: PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The Obesity Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-3027
Record Dates: First submitted 2019-06-03; First posted 2019-06-04 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Overweight and Obesity; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simple (Experimental): This arm uses a simplified form of dietary tracking that involves tracking only high-calorie, high-fat foods, in addition to the core behavioral smartphone-delivered intervention that consists of weighing, physical activity, goal setting, adaptive text messages, tailored weekly feedback, and lessons.
  Interventions: Behavioral: Simple
- Standard (Experimental): This arm uses standard calorie tracking, in addition to the core behavioral smartphone-delivered intervention that consists of weighing, physical activity, goal setting, adaptive text messages, tailored weekly feedback, and lessons.
  Interventions: Behavioral: Standard

INTERVENTIONS:
Behavioral: Simple — Participants have three daily goals (weighing, dietary goal, activity goal), will self-monitor (weigh on Wi-Fi enabled scale, use a simplified form of tracking only high-calorie, high-fat foods in the study smartphone app, wear Fitbit activity tracker), will receive 4-5 tailored text messages each week, and will view weekly tailored feedback and lessons in smartphone app.
  Arms: Simple
Behavioral: Standard — Participants have three daily goals (weighing, dietary goal, activity goal), will self-monitor (weigh on Wi-Fi enabled scale, track calorie intake, wear Fitbit activity tracker), will receive 4-5 tailored text messages each week, and will view weekly tailored feedback and lessons in smartphone app.
  Arms: Standard

SUMMARY:
The purpose of this study is to test the efficacy of an innovative 6-month smartphone-delivered intervention using simplified monitoring of dietary intake compared to a smartphone-delivered intervention with standard calorie monitoring among parents with overweight or obesity.

DETAILED DESCRIPTION:
This is a 6-month randomized controlled trial comparing the efficacy of two smartphone-based dietary and weight change interventions among 70 parent-child dyads with at least one child between the ages of 2 and 12 (70 adults and 70 children ages 2-12). One intervention group (Simple) will use a simplified, low-burden form of dietary tracking in the study smartphone application and the other group (Standard) will use standard calorie tracking. Components of both interventions include (1) setting personalized goals for weight, dietary intake, and daily activity (2) adaptive text message interventions based on behavior change techniques such as goal setting and in-the-moment progress feedback several times per week, (3) weekly tailored feedback updated in the study smartphone app, and (4) weekly lessons on the smartphone app. The primary objective is to promote weight loss in the parents, and the secondary objective is to determine if one or both interventions produce a ripple effect of parent dietary change onto dietary changes in the child.

ELIGIBILITY:
Inclusion Criteria (parent):

* Currently age 21-55.
* Body mass index (BMI) of 25-50 kg/m².
* Have one child between the ages of 2-12.
* Own an iPhone running at least iOS11 with a data and text messaging plan.
* Have the ability to read, write, and speak English.

Inclusion Criteria (child):

* Currently age 2-12.

Exclusion Criteria (parent):

* Lost more than 10 pounds in the last 6 months.
* Currently participating in another nutrition or weight loss program.
* Currently meeting exercise recommendations of 150 minutes per week of moderate-to-vigorous physical activity.
* Currently pregnant or breastfeeding, pregnant within the past 6 months, or planning to become pregnant within the next 6 months.
* Planning to relocate in the next 8 months.
* Will be out of town for 2 weeks or more in the next 8 months.
* Cannot attend two visits at the UNC Weight Research Program clinic.
* Pre-existing medical condition(s) that preclude adherence to an unsupervised exercise program, as determined by items endorsed on the PAR-Q (Physical Activity Readiness Questionnaire).
* Treatment of diabetes with insulin or oral medications that may cause hypoglycemia.
* History of clinically diagnosed eating disorder.
* Diagnosis of schizophrenia or bipolar disorder.
* Hospitalization for a psychiatric diagnosis within the last year.
* Report a past diagnosis of or current symptoms of alcohol or substance dependence.
* Another member of the household (family member or roommate) is a participant or staff member in this study.

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Percent weight loss: objective | Baseline, 6 Months
  Weight change from baseline to 6 months calculated as a percent from baseline weight.
Weight | Baseline, 6 Months
  Absolute weight change from baseline to 6 months.

SECONDARY OUTCOMES:
Dietary tracking adherence | from Baseline to 6 Months
  Number of days of complete dietary tracking summed over the 6-month study period.
Parent diet | Baseline, 6 Months
  Change in parent daily caloric intake as measured by 24-hour dietary recall from baseline to 6 months.
Child diet | Baseline, 6 Months
  Change in child daily caloric intake as measured by 24-hour dietary recall from baseline to 6 months.
Percent weight loss: WiFi scale | Baseline, 3 Months, 6 Months
  Weight change calculated as a percent from baseline weight (measured in kg), using official assessment weights taken from participants' study-provided WiFi-enabled weighing scale and transmitted via WiFi, from baseline to 3, and 6 months.
Child BMI-percentile | Baseline, 6 Months
  Change in child BMI-percentile using at-home measurements of child's weight (on parent WiFi-enabled scale) and height

OTHER OUTCOMES:
Minutes of moderate-to-vigorous physical activity | Baseline, 3 Months, 6 Months
  Change in minutes of moderate-to-vigorous physical activity as measured by the Paffenbarger Physical Activity Questionnaire, from baseline to 3, and 6 months. The PPAQ is a self-administered questionnaire that asks for a recall of physical activity over the previous 1 week. Participants report how many days and for how many minutes each day they engage in brisk walking, and report other exercise activities that week (non-occupational and non-household-related), including how many days and for how many minutes each time. Activities are assigned MET values according to the Compendium of Physical Activities, when are then used to classify activities as light moderate, or vigorous, and are also assigned energy expenditure amounts in kcal. These values are used to calculate total energy expenditure in kcal/week, as well as energy expenditure from and total minutes engaged in moderate-to-vigorous activities, measured in kcal/week and minutes/week, respectively.
Sedentary behavior | Baseline, 3 Months, 6 Months
  Change in sedentary behavior as measured by the self-administered Sedentary Behavior Questionnaire for Adults (SBQ), from baseline to 3, and 6 months. The SBQ asks about amount of sitting time on weekdays (8 items) and weekends (8 items), and are scored by summing up the total time spent in sedentary time (in hours) on weekdays and weekends, ranging from 0 hours to 6+ hours per day.
Physical food environment | Baseline, 3 Months, 6 Months
  Change in healthy and unhealthy foods offered in the home as measured by a physical food environment self-report questionnaire, from baseline to 3, and 6 months. There are 80 total items, 32 unhealthy items and 48 healthy items. Participants report whether each food/drink item is in the home or not (yes or no), and the items are summed for an unhealthy total and healthy total, and may also be used to total number of sugar-sweetened beverages/juice (out of 8 items), caloric beverages (15 items), fruits (17 items), vegetables (14 items), high-fat high-calorie items (20 items), and low-fat low-calorie items (14 items). Higher numbers indicate greater amounts of those types of food in the home.
Social food environment | Baseline, 3 Months, 6 Months
  Change in social food environment as measured by the Meals in our Household Questionnaire, from baseline to 3, and 6 months. This consists of 50 items across 6 subscales, summed to create a total score for each: structure of family meals (10 items, score range 0-40), problematic child mealtime behaviors (20 items, range 0-70), use of food as a reward (6 items, range 0-24), parental concern about child's diet (17 items, range 0-85), spousal stress related to child's mealtime behaviors (4 items, score range 4-20), and influence of child's food preferences on what other family members eat (3 items, range 2-14). Higher scores indicate higher instances of use of the scale in question (ex: greater structure of family meals, greater use of food as a reward, etc.).
Household food rules | Baseline, 3 Months, 6 Months
  Change in household food rules as measured by 12 items from the self-report Active Where Parent-Child Survey, from baseline to 3, and 6 months. The 12 items are summed to create a total score that ranges from 0-12, where higher scores indicate a greater number of food rules used.
Weight control self-efficacy | Baseline, 3 Months, 6 Months
  Change in weight control self-efficacy using the 20-item self-report Weight Efficacy Lifestyle Questionnaire, from baseline to 3, and 6 months. Items are rated on a scale of 0-9, and summed for a total score ranging from 0-180, with higher scores indicated greater self-efficacy.
Self-efficacy for exercise | Baseline, 3 Months, 6 Months
  Change in self-efficacy for exercise, as measured by the self-reported Self-Efficacy and Exercise Habits Survey, from baseline to 3, and 6 months. Responses for two subscales (Sticking to it - 8 items, Making time for exercise - 4 items) are averaged to yield a score from 1 to 5, with higher values representing higher self-efficacy for exercise.
Self-regulation | Baseline, 3 Months, 6 Months
  Change in self-regulation as measured by the 26-item self-report Eating Behavior Inventory, from baseline to 3, and 6 months. Scores range from 26-130, with higher scores indicating more use of positive eating behaviors.
Depressive symptoms | Baseline, 3 Months, 6 Months
  Change in depressive symptoms, as measured by the self-report 20-tem Center for Epidemiological Studies Depression Scale (CES-D), from baseline to 3, and 6 months. Scores range from 0-60, with higher scores indicating more depressive symptoms.
Stress | Baseline, 3 Months, 6 Months
  Change in stress, as measured by the self-report 10-item Perceived Stress scale, from baseline to 3 and 6 months. Scores range from 0-40, with higher scores indicating greater stress.

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Nezami, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882